CLINICAL TRIAL: NCT01625884
Title: Observational Study to Understand Patients' and Physicians' Attitudes to Statins in TurkeY
Acronym: STAY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CTR-XXX-2012/1
Record Dates: First submitted 2012-06-19; First posted 2012-06-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Hypercholesterolemia
Keywords: Statin; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In Turkey statin compliance is lower than EU countries. (EURIKA). We will assess the underlying causes of statin incompliance. The investigators will build patient and physician education programs to improve compliance in TURKEY. Our aim is to assess patients' and physicians' attitudes to statins by mean of HABIT Patient and Physician survey respectively.

DETAILED DESCRIPTION:
Observational study to understand patients' and physicians' attitudes to Statins in TurkeY

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent Female and/or male aged over 18 years,
* Diagnosis of hypercholesterolemia according to ICD-10 classification
* Receiving at least one prescription of one statin during the last 12 months and to be an outpatient.

Exclusion Criteria:

* Receiving statin at the time of admittance
* Patients unable to read and/or understand the study questionnaires
* Pregnant women,
* Patients participating in randomized clinical trials and patients included in this study once

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 18 years of age, diagnosed with hypercholesterolemia and prescribed with at least one statin irrespective of its type and/or dose. The inclusion period will last 6 months, on which consecutive patients attending the outpatient Family Physicians or Cardiologists office will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HABIT scores for the patients of the following questionnaire items (see description) | Participants will be questioned at visit one, visits will take part during 25 weeks of expected study period
  * Total score
  * Effectiveness of cholesterol-lowering medications
  * Association of high doses with adverse experiences
  * Risk of high cholesterol
  * Severity of high cholesterol
  * Frustration with the process of care
  * Difficulty in following advice / making changes
  * Doctor-patient communication
  * Communication about cholesterol
HABIT scores for the physicians of the following questionnaire items (see description) | Participants will be questioned at visit one, visits will take part during 25 weeks of expected study period
  * Total score
  * Effectiveness of statins
  * Patients view titration negatively
  * Risk associated with higher doses
  * Close enough to goal
  * Urgency of getting to goal
  * Utility of diet and exercise
  * Time and resources to counsel patients
  * Physician self-efficacy in treating patients to goal

SECONDARY OUTCOMES:
Socio-demographics terms | Participants will be questioned at visit one, visits will take part during 25 weeks of expected study period
  * Age
  * Sex
  * Smoking habits
  * Educational level
  * Professional status
  * Place of residence
  * Income level
  * Healthcare insurance level
Clinical characteristics | Participants will be questioned at visit one, visits will take part during 25 weeks of expected study period
  * Date of diagnosis
  * Current disease status: Physical examination results (vital signs and anthropometric measurements)
  * Cardiovascular risk factors
  * Relevant co-morbidities
  * Cholesterol levels (LDL-C) at inclusion (if available)
  * Number of hospitalizations during the last 12 months
  * Duration of statin use in the past year
Clinical characteristics (continuation) | Participants will be questioned at visit one, visits will take part during 25 weeks of expected study period
  * List of poor compliance (discontinuation) causes in the past one year
  * Treatment discontinuation (statins), reported causes
  * Time to discontinuation of statin therapy (in early stage/medium term/long term)
  * Change in lipid levels and other laboratory findings (i.e. hepatic and muscle enzymes) during statin use (before, during and after discontinuation of statin therapy)
  * List of alternative drug and non-drug therapies received after discontinuation of statin and number (%) of patients who switched to those alternative therapies
  * Concomitant treatments

CONTACTS AND LOCATIONS:
Overall Officials: Mujgan Ates, DR, Study Director — AZ MC Turkey; Ramazan Ozdemir, PROF.DR., Principal Investigator — Inonu University Faculty of Medicine, Cardiology Department
Locations (10):
- Turkey (Türkiye) (10):
  - Research Site, Ankara
  - Research name, Aydin
  - Research Site, Diyarbakır
  - Research Site, Hatay
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, K. Maras
  - Research Site, Kayseri
  - Research Site, Malatya
  - Research Site, Manisa

REFERENCES:
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; Coordinating Committee of the National Cholesterol Education Program. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III Guidelines. J Am Coll Cardiol. 2004 Aug 4;44(3):720-32. doi: 10.1016/j.jacc.2004.07.001. PMID 15358046
- [Background] Pearson TA, Laurora I, Chu H, Kafonek S. The lipid treatment assessment project (L-TAP): a multicenter survey to evaluate the percentages of dyslipidemic patients receiving lipid-lowering therapy and achieving low-density lipoprotein cholesterol goals. Arch Intern Med. 2000 Feb 28;160(4):459-67. doi: 10.1001/archinte.160.4.459. PMID 10695686
- [Background] Ertas FS. [Statins with a perspective of lifelong therapy]. Turk Kardiyol Dern Ars. 2009 Mar;37 Suppl 2:29-36. Turkish. PMID 19404048
- [Background] Tokgozoglu L, Kaya EB, Erol C, Ergene O; EUROASPIRE III Turkey Study Group. [EUROASPIRE III: a comparison between Turkey and Europe]. Turk Kardiyol Dern Ars. 2010 Apr;38(3):164-72. Turkish. PMID 20675993
- [Background] Ford I, Murray H, Packard CJ, Shepherd J, Macfarlane PW, Cobbe SM; West of Scotland Coronary Prevention Study Group. Long-term follow-up of the West of Scotland Coronary Prevention Study. N Engl J Med. 2007 Oct 11;357(15):1477-86. doi: 10.1056/NEJMoa065994. PMID 17928595
- [Background] Benner JS, Glynn RJ, Mogun H, Neumann PJ, Weinstein MC, Avorn J. Long-term persistence in use of statin therapy in elderly patients. JAMA. 2002 Jul 24-31;288(4):455-61. doi: 10.1001/jama.288.4.455. PMID 12132975
- [Background] Ho PM, Magid DJ, Shetterly SM, Olson KL, Maddox TM, Peterson PN, Masoudi FA, Rumsfeld JS. Medication nonadherence is associated with a broad range of adverse outcomes in patients with coronary artery disease. Am Heart J. 2008 Apr;155(4):772-9. doi: 10.1016/j.ahj.2007.12.011. PMID 18371492
- [Background] Shah ND, Dunlay SM, Ting HH, Montori VM, Thomas RJ, Wagie AE, Roger VL. Long-term medication adherence after myocardial infarction: experience of a community. Am J Med. 2009 Oct;122(10):961.e7-13. doi: 10.1016/j.amjmed.2008.12.021. Epub 2009 Jun 26. PMID 19560749
- [Background] Glader EL, Sjolander M, Eriksson M, Lundberg M. Persistent use of secondary preventive drugs declines rapidly during the first 2 years after stroke. Stroke. 2010 Feb;41(2):397-401. doi: 10.1161/STROKEAHA.109.566950. Epub 2010 Jan 14. PMID 20075360
- [Background] Lardizabal JA, Deedwania PC. Benefits of statin therapy and compliance in high risk cardiovascular patients. Vasc Health Risk Manag. 2010 Oct 5;6:843-53. doi: 10.2147/VHRM.S9474. PMID 20957130
- [Background] Yang Y, Thumula V, Pace PF, Banahan BF 3rd, Wilkin NE, Lobb WB. Predictors of medication nonadherence among patients with diabetes in Medicare Part D programs: a retrospective cohort study. Clin Ther. 2009 Oct;31(10):2178-88; discussion 2150-1. doi: 10.1016/j.clinthera.2009.10.002. PMID 19922889
- [Background] Chan DC, Shrank WH, Cutler D, Jan S, Fischer MA, Liu J, Avorn J, Solomon D, Brookhart MA, Choudhry NK. Patient, physician, and payment predictors of statin adherence. Med Care. 2010 Mar;48(3):196-202. doi: 10.1097/MLR.0b013e3181c132ad. PMID 19890219
- [Background] Foley KA, Vasey J, Berra K, Alexander CM, Markson LE. The Hyperlipidemia: Attitudes and Beliefs in Treatment (HABIT) survey for patients: results of a validation study. J Cardiovasc Nurs. 2005 Jan-Feb;20(1):35-42. doi: 10.1097/00005082-200501000-00008. PMID 15632811
- [Background] Foley KA, Vasey J, Alexander CM, Markson LE. Development and validation of the hyperlipidemia: attitudes and beliefs in treatment (HABIT) survey for physicians. J Gen Intern Med. 2003 Dec;18(12):984-90. doi: 10.1111/j.1525-1497.2003.30114.x. PMID 14687256
- See also: NIS-CTR-XXX-2012/1 Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=849&filename=NIS-CTR-XXX-2012_1.pdf